CLINICAL TRIAL: NCT00405301
Title: Study of Safety and Efficacy of Different Regimes of Reintroduction of Anti-TB Drugs in Antituberculosis Treatment Induced Hepatotoxicity
Brief Title: Study of Safety and Efficacy of Different Regimes of Reintroduction of Anti-TB Drugs in Anti-TB Drugs Induced Liver Damage
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: All India Institute of Medical Sciences (Other)
Responsible Party: Principal Investigator, S.K.SHARMA, Professor and Head, All India Institute of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AIIMS/MED/2006/10
Record Dates: First submitted 2006-11-27; First posted 2006-11-30 (Estimated); Last update posted 2012-02-16 (Estimated); Status verified 2012-02

CONDITIONS: Drug Induced Hepatotoxicity; Tuberculosis
Keywords: Tuberculosis; Drug Induced Hepatotoxicity; Anti-tuberculosis drugs; India
MeSH Terms: conditions — Chemical and Drug Induced Liver Injury; Tuberculosis | interventions — Pyrazinamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm 1 (Other): Arm 1: will receive Isoniazide(5mg/kg/day), Rifampicin(10mg/kg/day) and Pyrazinamide(25mg/kg/day) in full doses on day 1 and continued further
  Interventions: Drug: Rifampicin(max dose 10 mg/kg/day), Isoniazide (max dose 5 mg/kg/day) and Pyrazinamide (max dose 25 mg/kg/day)
- Arm 2 (Other): Arm 2 : will receive Rifampicin(10mg/kg/day) in full dose on day 1 and continued, Isoniazide(5mg/kg/day)in full dose on day 8 and continued, Pyrazinamide(25mg/kg/day)on day 15 and continued
  Interventions: Drug: Rifampicin(max dose 10 mg/kg/day), Isoniazide (max dose 5 mg/kg/day) and Pyrazinamide (max dose 25 mg/kg/day)
- Arm 3 (Other): Arm 3 will receive 100 mg/day of Isoniazide on day 1 which is gradually increased to maximum dose (5mg/kg/day) by day 4 and continued. Rifampicin is introduced on day 8 in a dose of 150 mg/day which is gradually increased to maximum dose (10mg/kg/day) by day 11 and continued. Pyrazinamide is introduced on day 15 in a dose of 500mg/day which is gradually increased to maximum dose (25mg/kg/day) by day 18 and continued.
  Interventions: Drug: Rifampicin(max dose 10 mg/kg/day), Isoniazide (max dose 5 mg/kg/day) and Pyrazinamide (max dose 25 mg/kg/day)

INTERVENTIONS:
Drug: Rifampicin(max dose 10 mg/kg/day), Isoniazide (max dose 5 mg/kg/day) and Pyrazinamide (max dose 25 mg/kg/day) — Patients who develop ATT drug induced hepatotoxicity will be divided into 3 arms .Arm 1,2,3 will be given drugs as described in detailed description of the title.

SUMMARY:
Purpose of the study is to evaluate the safety and efficacy of different re-introduction regimens in anti-TB drug induced liver damage. There is no consensus how best to treat such patients who developed drug induced liver damage.

DETAILED DESCRIPTION:
Tuberculosis continues to be a major health problem in both the developing and developed countries because of its resurgence in the immunosuppressed patients. Short course chemotherapy containing isoniazid, rifampicin and pyrazinamide has proved to be highly effective in the treatment of tuberculosis. One of its adverse effect is liver damage which is the most common side effect leading to interruption of therapy.

There is lack of consensus guidelines for treatment of anti-TB drug induced liver damage Whether the re-introduction should take place with all the drugs given together in full doses (which reduces the chance of resistance and cost to the patient) or in a phased manner. There is lack of studies which compared different regimens of re-introduction of anti-TB drugs.

In this study, we will study three regimes of re-introduction of hepatotoxic anti-tuberculosis drugs (Rifampicin, Isoniazide, Pyrazinamide). These are potent anti-tuberculosis medications and need to be restarted in patients who developed liver toxicities attributed to these medications and became normal when these medicines were stopped. At the time of re-introduction the patients will be randomized in 3 groups.

* First group will receive Isoniazide(5mg/kg/day), Rifampicin(10mg/kg/day) and Pyrazinamide(25mg/kg/day) in full doses on day 1 and continued further.
* second group will receive Rifampicin(10mg/kg/day) in full dose on day 1 and continued, Isoniazide(5mg/kg/day)in full dose on day 8 and continued, Pyrazinamide(25mg/kg/day)on day 15 and continued.
* Third group will receive 100 mg/day of Isoniazide on day 1 which is gradually increased to maximum dose (5mg/kg/day) by day 4 and continued. Rifampicin is introduced on day 8 in a dose of 150 mg/day which is gradually increased to maximum dose (10mg/kg/day) by day 11 and continued. Pyrazinamide is introduced on day 15 in a dose of 500mg/day which is gradually increased to maximum dose (25mg/kg/day) by day 18 and continued.

All the three groups will be monitored for three months by analyzing weekly liver function tests. Any difference in the morbidity, deranged liver function or any other adverse effects will be monitored and treated appropriately.

ELIGIBILITY:
Inclusion Criteria:

* A rise of five times the upper limit of the normal levels (50 IU/L) of serum aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT)
* A rise in the level of serum total bilirubin level > 1.5mg/dl
* Any increase in serum AST and or ALT above pretreatment values together with anorexia, nausea, vomiting and jaundice
* Absence of serological evidence of infection with hepatitis viruses A,B,C,or E
* Normalization of liver function tests after withdrawal of antituberculosis drugs For diagnosis of anti-TB drugs induced hepatitis, criteria 1 or 2 or 3 should be present along with criteria 4 and 5.

Exclusion Criteria:

* Patients with serological evidence of acute viral hepatitis A,B,C,or E and carriers for HBV & HCV
* Age < 15 year and age > 65 years
* HIV positive patients
* Presence of chronic liver disease or cirrhosis
* Co-administration of other potential hepatotoxic drugs (methotrexate, phenytoin, valproate)
* Chronic alcoholics who consume > 48 g of alcohol/day for at least one year
* Pregnant women
* Subjects not giving consent

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 175 (Actual)
Dates: Start 2006-12; Primary Completion 2008-06 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
To compare the safety of different regimens of re-introduction of anti-TB drugs in drug induced liver damage. | 24 months

SECONDARY OUTCOMES:
To study the predictors of recurrence of drug induced liver damage | 24 months
To study the risk factors for development of drug induced liver injury | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Surendra K Sharma, MD, PhD, Principal Investigator — All India Institute of Medical Sciences
Locations (2):
- India (2):
  - Sri Venkateswara Institute of Medical Sciences, Tirupati, Andhra Pradesh
  - All India Institute of Medical Sciences, New Delhi, National Capital Territory of Delhi

REFERENCES:
- [Background] Tahaoglu K, Atac G, Sevim T, Tarun T, Yazicioglu O, Horzum G, Gemci I, Ongel A, Kapakli N, Aksoy E. The management of anti-tuberculosis drug-induced hepatotoxicity. Int J Tuberc Lung Dis. 2001 Jan;5(1):65-9. PMID 11263519
- [Background] Singh J, Garg PK, Tandon RK. Hepatotoxicity due to antituberculosis therapy. Clinical profile and reintroduction of therapy. J Clin Gastroenterol. 1996 Apr;22(3):211-4. doi: 10.1097/00004836-199604000-00012. PMID 8724260
- [Background] Singh J, Arora A, Garg PK, Thakur VS, Pande JN, Tandon RK. Antituberculosis treatment-induced hepatotoxicity: role of predictive factors. Postgrad Med J. 1995 Jun;71(836):359-62. doi: 10.1136/pgmj.71.836.359. PMID 7644398
- [Background] Sharma SK, Balamurugan A, Saha PK, Pandey RM, Mehra NK. Evaluation of clinical and immunogenetic risk factors for the development of hepatotoxicity during antituberculosis treatment. Am J Respir Crit Care Med. 2002 Oct 1;166(7):916-9. doi: 10.1164/rccm.2108091. PMID 12359646
- [Background] Sharma SK. Antituberculosis drugs and hepatotoxicity. Infect Genet Evol. 2004 Jun;4(2):167-70. doi: 10.1016/j.meegid.2003.01.001. No abstract available. PMID 15157635
- [Derived] Sharma SK, Singla R, Sarda P, Mohan A, Makharia G, Jayaswal A, Sreenivas V, Singh S. Safety of 3 different reintroduction regimens of antituberculosis drugs after development of antituberculosis treatment-induced hepatotoxicity. Clin Infect Dis. 2010 Mar 15;50(6):833-9. doi: 10.1086/650576. PMID 20156055